CLINICAL TRIAL: NCT06441565
Title: Fruquintinib Plus Arterial Infusion Therapy With Hepatic FOLFOX for Refractory Colorectal Cancer: The FAITH Randomized Clinical Trial
Brief Title: Fruquintinib With or Without HAI-FOLFOX for Refractory Colorectal Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuhong Li, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAITH-CRC
Record Dates: First submitted 2024-05-24; First posted 2024-06-04 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Hepatic Arterial Infusion Chemotherapy; Randomized Clinical Study; Progression Free Surivival; Safety Profile
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to either the fruquintinib monotherapy group (control group) or the fruquintinib plus HAI-FOLFOX treatment group (experimental group)
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fruquintinib monotherapy group (control group) (Active Comparator): Participants in the fruquintinib monotherapy group will undergo a treatment cycle every 4 weeks, taking 5 mg orally once daily for 3 weeks, followed by a 1-week break.
  Interventions: Drug: Fruquintinib
- Fruquintinib plus HAI-FOLFOX treatment group (experimental group) (Experimental): The experimental group will receive fruquintinib plus HAI-FOLFOX, with HAI-FOLFOX given every 2 weeks
  Interventions: Drug: Fruquintinib; Drug: Fluorouracil; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Fruquintinib — A treatment cycle of 4 weeks, with 5 mg orally once daily for 3 weeks, followed by a 1-week break
  Other Names: Fruzaqla
Drug: Fluorouracil — 2.8 g/m² (400mg bolus + 2.4g/m² continuous infusion) given every 2 weeks through hepatic arterial infusion
  Other Names: 5-FU
  Arms: Fruquintinib plus HAI-FOLFOX treatment group (experimental group)
Drug: Oxaliplatin — 85 mg/m² given every 2 weeks through hepatic arterial infusion
  Other Names: L01XA03
  Arms: Fruquintinib plus HAI-FOLFOX treatment group (experimental group)

SUMMARY:
The objective of this clinical trial is to evaluate the efficacy and safety of combining fruquintinib with hepatic artery infusion (HAI)-FOLFOX in the treatment of refractory colorectal cancer with liver metastasis.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer globally, accounting for approximately 10% of all cancer cases, and is the second leading cause of cancer-related deaths worldwide. Significant advancements have been made in treating metastatic colorectal cancer (mCRC) over the past two decades, primarily due to continuous improvements in first-line treatment regimens. However, treatment options are relatively limited for patients with mCRC who do not respond to standard first-line treatments or who develop chemotherapy resistance. Approved second-line treatments include regorafenib, fruquintinib, and TAS-102, but their reported efficacy and overall survival (OS) rates are not ideal.

Fruquintinib is a novel small-molecule anticancer drug classified as a quinazoline, acting as a potent and highly selective inhibitor of vascular endothelial growth factor receptor (VEGFR) tyrosine kinase. Preclinical and clinical studies conducted in China and the United States have demonstrated significant anticancer activity of fruquintinib in solid tumors. The prospective randomized controlled clinical study FRESCO-2 showed that fruquintinib significantly improved median OS (7.4 months vs. 4.8 months; P < 0.001) and median progression-free survival (PFS) (3.7 months vs. 1.8 months; P < 0.001) compared to the placebo group. These results are consistent with previous FRESCO study findings. Although these studies provide strong evidence for fruquintinib in treating refractory mCRC patients, the overall improvement in survival is limited, with a 6-month PFS rate of only about 20% (FRESCO: 19.3%, FRESCO-2: 22.7%). Thus, there is a need for new second-line treatment options to further enhance efficacy and survival in refractory mCRC patients.

Recent studies have shown that combining fruquintinib with paclitaxel as a second-line therapy demonstrates good efficacy and safety in advanced gastric cancer patients. Additionally, fruquintinib combined with sintilimab has shown some antitumor activity, particularly in mCRC patients with pMMR status. Therefore, combining fruquintinib with other anticancer drugs might offer a new treatment direction for refractory mCRC.

Liver metastasis is the most common form of metastasis in colorectal cancer. Normal liver tissue primarily receives blood supply from the portal vein, while colorectal cancer liver metastases mainly receive blood from the hepatic artery. This dual blood supply characteristic has led to the development of hepatic artery infusion (HAI), a treatment method delivering high concentrations of chemotherapy drugs directly to liver metastases, minimizing toxicity to normal liver tissue and surrounding organs. For mCRC patients with chemotherapy resistance and liver-dominant metastasis, treatments such as yttrium-90 resin microsphere selective internal radiation therapy (Y-90 SIRT) are recommended by NCCN guidelines, although Y-90 SIRT is not yet widely available domestically. Fluorouracil (5-FU) and floxuridine (FUDR) are the most commonly used drugs for hepatic artery infusion chemotherapy (HAIC), with high first-pass metabolism rates and short half-lives, suitable for HAI. Studies have reported that HAIC combined with systemic chemotherapy shows high efficacy (76%) and a conversion surgery rate of 47% in mCRC patients who have undergone multiple lines of treatment. Cercek et al. found that mCRC patients resistant to at least three standard systemic treatments (n = 57) benefited from HAI-FUDR, with partial response (PR) and stable disease (SD) rates of 33% and 54%, respectively. However, many countries, including China, no longer produce FUDR injections, necessitating the search for alternative drugs or combinations for HAIC.

Compared to systemic oxaliplatin chemotherapy, hepatic artery infusion chemotherapy with oxaliplatin has a high hepatic extraction rate of 0.47 and good safety. A phase II clinical study using oxaliplatin HAIC combined with intravenous 5-FU as first-line treatment showed an objective response rate (ORR) of 64% and a median OS of 27 months in patients with unresectable CRLM. Another study by the same team found that oxaliplatin HAIC had a disease control rate of 87% (n = 39) in CRLM patients who had previously received FOLFIRI or FOLFOX treatments, with 62% achieving partial response, suggesting that oxaliplatin-based HAIC could overcome resistance to previous oxaliplatin-containing systemic therapies. Due to these promising results, several prospective randomized clinical studies are currently underway, such as the phase II SULTAN study investigating oxaliplatin HAIC combined with systemic FOLFIRI as salvage therapy in patients with unresectable localized mCRC after systemic chemotherapy induction. Recent retrospective studies and randomized clinical trials have confirmed that HAI-FOLFOX alone or in combination with other drugs significantly improves the prognosis of patients with advanced hepatocellular carcinoma. Our previous retrospective analysis of 21 patients with recurrent, unresectable CRLM after multiple lines of treatment, who received oxaliplatin + 5-FU (FOLFOX) or FUDR HAIC with or without systemic chemotherapy, showed an ORR of 28.6%, with 7 patients successfully undergoing conversion surgery. The median PFS was 6.3 months, with a 6-month PFS rate of 61.9%. However, due to the limited sample size and retrospective design of our study, caution is needed when generalizing these results.

To address the limitations of previous studies and provide more robust evidence, this prospective randomized clinical study will investigate the synergistic effects of combining fruquintinib with HAI-FOLFOX. The aim is to determine whether this combination improves the efficacy in CRLM patients who have progressed after standard systemic chemotherapy compared to fruquintinib monotherapy. By systematically observing a larger patient sample, we hope to understand the potential advantages of this treatment regimen in improving PFS, ORR, and OS. This prospective study will provide valuable insights into the potential clinical benefits of fruquintinib combined with HAI-FOLFOX, paving the way for new treatment strategies and advancing personalized treatment for patients with refractory metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years.
* Histologically confirmed colorectal adenocarcinoma.
* Radiologically or pathologically confirmed liver metastasis.
* At least one measurable lesion (per RECIST v1.1 criteria).
* No extrahepatic metastasis confirmed by CT, MRI, or PET/CT (if necessary). Patients with minimal extrahepatic metastatic burden (defined as the presence of lung metastasis and/or lymph node metastasis with lung lesion diameter not exceeding 1 cm, and lymph node metastasis with the longest diameter less than 2 cm) can be included.
* Disease progression within 3 months or intolerance to standard treatment with fluoropyrimidine, irinotecan, oxaliplatin combined with targeted therapy (including bevacizumab and cetuximab (RAS/BRAF wild-type)), with previous oxaliplatin-induced neurotoxicity < Grade 2.
* Normal hematologic function (platelets >90×10^9/L; white blood cells >3×10^9/L; neutrophils >1.5×10^9/L).
* Serum bilirubin ≤1.5 times the upper limit of normal (ULN), transaminases ≤5 times ULN, alkaline phosphatase ≤2.5 times ULN, no ascites, coagulation function: prothrombin time (PT) ≤1.5 ULN; international normalized ratio (INR) ≤1.5 ULN; activated partial thromboplastin time (APTT) ≤1.5 ULN, albumin ≥35 g/L.
* Child-Pugh grade A liver function.
* Serum creatinine less than ULN, or calculated creatinine clearance >50 ml/min (using Cockcroft-Gault formula).
* ECOG performance status 0-1.
* Expected survival >3 months.
* Signed written informed consent.
* Willing and able to undergo follow-up until death or study completion/termination.

Exclusion Criteria:

* Severe arterial embolism.
* Bleeding tendency or coagulation disorders.
* Hypertensive crisis or hypertensive encephalopathy.
* Severe uncontrolled systemic complications such as infection or diabetes.
* Clinically significant cardiovascular diseases such as cerebrovascular accident (within 6 months prior to enrollment), myocardial infarction (within 6 months prior to enrollment), uncontrolled hypertension despite appropriate medical therapy, unstable angina, congestive heart failure (NYHA Class 2-4), or arrhythmias requiring medication.
* History or physical examination indicative of central nervous system diseases (e.g., primary brain tumors, uncontrolled seizures, any history of brain metastasis or stroke).
* Other malignancies within the past 5 years (except for radically treated basal cell carcinoma of the skin and/or carcinoma in situ of the cervix).
* Received any investigational drug treatment within 28 days prior to the study.
* Residual toxicity from previous chemotherapy (excluding alopecia), such as peripheral neuropathy ≥ Grade 2 (NCI CTCAE v5.0), if considering an oxaliplatin-containing regimen.
* Allergy to any of the study drugs.
* Pregnant or breastfeeding women.
* Women of childbearing potential not using or refusing to use effective non-hormonal contraception (intrauterine device, barrier method combined with spermicide, or sterilization) or men with reproductive potential.
* Inability or unwillingness to comply with the study protocol.
* Presence of any other diseases, functional impairment due to metastatic lesions, or findings on physical examination suggesting a contraindication to the use of the study drugs or putting the participant at high risk for treatment-related complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival | Assessed 6 months following treatment initiation
  The proportion of patients who remain alive and whose disease does not progress over a period of six months after starting treatment

SECONDARY OUTCOMES:
Liver Lesion Progression-Free Survival | Assessed throughout the study duration (5 years)
  Duration of time during which liver metastases remain stable without progression.
Extrahepatic Lesion Progression-Free Survival (PFS) | Assessed throughout the study duration (5 years)
  Duration of time during which metastases outside the liver remain stable without progression.
Liver Lesion Objective Response Rate | Assessed throughout the study duration (5 years)
  Proportion of patients achieving partial or complete response in liver metastases per RECIST criteria.
Extrahepatic Lesion Objective Response Rate (ORR) | Assessed throughout the study duration (5 years)
  Proportion of patients achieving partial or complete response in extrahepatic metastases per RECIST criteria.
Overall Survival | Assessed throughout the study duration (5 years)
  Time from treatment initiation to death from any cause or censored due to loss to follow up
Adverse events (catheter related and chemotherapy related) | Assessed throughout the study duration (5 years)
  Assessment of adverse events and their severity according to NCI CTCAE version 5.0 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Data and materials used in this study can be made available following study completion upon reasonable request to the corresponding author, subject to ethical and legal considerations and applicable data-sharing agreements.